CLINICAL TRIAL: NCT06170125
Title: A Multicenter, Non-interventional, Observational Clinical Trial to Assess the Quality of Life in Patients With ChRonic ObstructIve Pulmonary Disease Who Require Tiotropium as additiOnal treatmeNt.
Brief Title: QualiTy of Life Evaluation in Patients With ChRonic ObstructIve Pulmonary Disease Who Require Tiotropium as additiOnal treatmeNt.
Acronym: TRITON
Status: Not yet recruiting | Type: Observational
Sponsor: Elpen Pharmaceutical Co. Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 2023-TIO-EL-187
Record Dates: First submitted 2023-11-28; First posted 2023-12-14 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-01

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Tiotropium treated patients — Patients who are not satisfied with their COPD treatment and will be on additional tiotropium scheme.

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is a complex, heterogeneous disease usually with a decline lung function and worsening symptoms; hence, both forced expiratory volume in 1 s (FEV1; lung function) and validated patient-reported outcomes (PROs) are used in clinical trials to assess disease severity and response to treatment.

The PROs are different in terms of their scope of assessment and in the information that they capture. PRO questionnaires such as the Baseline Dyspnoea Index (BDI), Transition Dyspnoea Index (TDI) and modified Medical Research Council (mMRC) dyspnoea scale are used to assess dyspnoea, whereas the Clinical COPD Questionnaire (CCQ), COPD Assessment Test (CAT) and St George's Respiratory Questionnaire (SGRQ) are commonly used to assess patients' health status .

Furthermore, the mMRC scale is unidirectional and minimally responsive to treatment interventions, while the BDI, TDI, CAT, CCQ and SGRQ (approved by the USA Food and Drug Administration) are multidirectional.

DETAILED DESCRIPTION:
With the availability of numerous PROs, it is important to understand which provide a better evaluation of patients' health status and demonstrate responses to treatment. Even when PROs evaluate the same parameter, e.g. dyspnoea, they may not always capture a uniform response. Hence, it would be useful to examine if the PROs correlate with each other and whether any specific PROs better reflect treatment benefit (as expressed by minimal clinically important differences (MCIDs)) than the others. Furthermore, understanding the relationship between the PROs and lung function (FEV1) may provide insights into whether a change in lung function translates to a change perceptible by the patients (assessed through PROs).

Tiotropium is a potent, long-acting, selective anticholinergic bronchodilator. Treatment with tiotropium produces sustained improvements in lung function, particularly FEV1 (peak, trough, average, and area under the curve) compared with either placebo or ipratropium in patients with moderate to severe COPD. Preliminary evidence suggests that treatment with tiotropium may slow the rate of decline in FEV1, but this finding awaits confirmation. Tiotropium reduces lung hyperinflation, with associated improvements in exercise capacity. Tiotropium, compared with either placebo or ipratropium, improves a variety of patient-centered outcomes, including subjective dyspnea ratings and Health Related Quality of Life (HRQL) scores. Tiotropium reduces the frequency of COPD exacerbations and of hospitalizations due to exacerbations, but has not been shown to reduce all-cause mortality. Compared with the long-acting bronchodilators, tiotropium provides incrementally better bronchodilation, but it is not clearly superior in terms of patient-centered outcomes. Tiotropium has a good safety profile; however patients with severe cardiac disease, bladder outlet obstruction, or narrow angle glaucoma were excluded from all studies.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (≥40 years old) with a diagnosis of Chronic Respiratory Pulmonary Disease (COPD).
2. Patients who were treated with Inhaled Corticosteroid (ICS)/LABA, LABA/LAMA with a LABA or ICS/LABA or were not receiving long-acting bronchodilators (LABA or LAMA) for COPD and required addition of tiotropium from 1 to 7 days before the start of the study.
3. Patients who are able to provide informed consent and follow study procedures and requirements.

Exclusion Criteria:

1. According to the contraindications of the product's Summary of Product Characteristics.
2. Patients receiving LAMA monotherapy prior to study entry.

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients patients (≥40 years old) with a diagnosis of Chronic Respiratory Pulmonary Disease (COPD) who were treated with ICS/LABA, LABA/LAMA with a LABA or ICS/LABA or were not receiving long-acting bronchodilators (LABA or LAMA) for COPD and required addition of tiotropium from 1 to 7 days before the start of the study.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Quality of Life assesment | 6 months
  Change in Clinical COPD Questionnaire (CCQ)

SECONDARY OUTCOMES:
Dyspnea assesment | 6 months
  Change in Baseline Dyspnoea Index, BDI at baseline and Transition Dyspnoea Index, TDI between study visits and after 6 months treatment.
COPD Assessment Test | 6 months
  Change in CAT (COPD Assessment Test) between study visits and after 6 months of treatment.
FEV1 % predicted measurement | 6 months
  Change in FEV1% predicted and other spirometric parameters (FEV1, FVC, FEV1/FVC) during study visits and after 6 months of tiotropium treatment
Feeling of Satisfaction with Inhaler (FSI-10) questionnaire | 6 months
  Change in FSI-10 questionnaire for patients satisfaction after 6 months of tiotropium treatment.
Exacerbations | 6 months
  Report of number of median exacerbations that will be appeared during 6 months of tiotropium treatment
Adverse Events | 6 months
  Report the number of Adverse Events during study period

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kostikas K, Greulich T, Mackay AJ, Lossi NS, Aalamian-Mattheis M, Nunez X, Pagano VA, Patalano F, Clemens A, Vogelmeier CF. Treatment response in COPD: does FEV1 say it all? A post hoc analysis of the CRYSTAL study. ERJ Open Res. 2019 Feb 25;5(1):00243-2018. doi: 10.1183/23120541.00243-2018. eCollection 2019 Feb. PMID 30815470
- [Background] Kostikas K, Mackay AJ, Vogelmeier CF, Frent SM, Gupta P, Banerji D, Patalano F, Pfister PJ, Wedzicha JA. Early Clinically Important Improvement (ECII) and Exacerbation Outcomes in COPD Patients. Int J Chron Obstruct Pulmon Dis. 2020 Jul 28;15:1831-1838. doi: 10.2147/COPD.S247966. eCollection 2020. PMID 32884253
- [Background] Anzueto A, Miravitlles M. Tiotropium in chronic obstructive pulmonary disease - a review of clinical development. Respir Res. 2020 Jul 29;21(1):199. doi: 10.1186/s12931-020-01407-y. PMID 32727455